CLINICAL TRIAL: NCT04522362
Title: Modeling Stress-precipitated Vaping Behavior Among E-Cigarette Users
Brief Title: Modeling Stress-precipitated Vaping Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: University of Vermont (Other)
Responsible Party: Principal Investigator, Irene Pericot-valverde, Research Assistant Professor, Clemson University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 17-0498
Record Dates: First submitted 2020-08-13; First posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control task- (Sham Comparator): The Control Task was implemented to ensure the specificity of the psychological stress effects had on study outcomes. Therefore, the Control Task had a similar procedure and the same duration of the TSST, lacking except for only the psychologically stressful component. The control task consisted of (a) Participants had a 5-min a preparation section and anticipation phase (5 min ), (b) a reading task where they had to. Then, all participants had to be read a simple text in a low voice (5 min), and (c) an arithmetic section where they were asked to perform an easy mathematical calculation (5 mins).
  Interventions: Other: Control task and Trier Social Stress Task
- Experimental Task- Trier Social Stress Task (Experimental): The Trier Social Stress Task (TSST) is a standardized, 15-minute laboratory task designed to induce psychological stress in laboratory settings (Kirschbaum, Pirke, & Hellhammer, 1993). The TSST consists of three continuously successive phases: (a) an anticipation period (5 min); (b) a free speech task (5 min); and (c) a mental arithmetic task (5 min). As is standard in the TSST procedure, participants were told by a research staff member that they would provide a brief speech about "their dream job" in front of a critical audience. At the end of the speech, a member of the audience instructed the participant to conduct serial subtractions as accurately and quickly as possible.
  Interventions: Other: Control task and Trier Social Stress Task

INTERVENTIONS:
Other: Control task and Trier Social Stress Task — Same as Arm

SUMMARY:
The primary aims of this pilot study were to (1) initially validate the applicability of a human laboratory model of relapse initially developed for smokers to e-cigarette users; (2) to use this human laboratory model of lapse behavior to examine the effects of acute psychological stress on vaping-lapse behavior among adults who are experienced, e-cigarette users.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* e-cigarette users
* using ≥1 mL of e-cigarette liquid per day with a nicotine concentration of ≥3mg/ml
* had used an e-cigarette for at least three months

Exclusion Criteria:

* Current smokers
* Psychiatric or medical condition based
* Using a prescription medication other than birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
latency to initiate ad-lib vaping session (in minutes) | During the two laboratory sessions which occur within 1 week after screening/baseline.
  Time to vaping during the vaping delay task. Range of time delay is 0 minutes to 50 minutes.
number of puffs purchased and consumed during the self-administration period | During the two laboratory sessions which occur within 1 week after screening/baseline
  Number of e-cigarette uses purchased during the self-administration phase of the vaping delay task. Range of puffs is 0 to 20.

SECONDARY OUTCOMES:
Craving | The VAS will be collected at each laboratory session (within 1 week after screening/baseline) 5 times: baseline (pre task), post task (+15 minutes), decision to smoke (+20 minutes), +30 minutes smoking ab-lib, and +60 minutes during smoking ab-lib
  Craving was measured using a visual analogue scale (VAS) asking "How much do you crave an e-cigarette right now?" with possible responses ranging from 0 (not at all) to 100 (extremely).
Stress | The VAS will be collected at each laboratory session (within 1 week after screening/baseline) 5 times: baseline (pre task), post task (+15 minutes), decision to smoke (+20 minutes), +30 minutes smoking ab-lib, and +60 minutes during smoking ab-lib
  Stress was measured using a visual analogue scale (VAS) asking: "How stressed or anxious do you feel right now?" with possible responses ranging from 0 (not at all) to 100 (extremely).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pericot-Valverde I, Yoon JH, Byrne KA, Heo M, Niu J, Litwin AH, Gaalema DE. Effects of short-term nicotine deprivation on delay discounting among young, experienced, exclusive ENDS users: An initial study. Exp Clin Psychopharmacol. 2023 Jun;31(3):724-732. doi: 10.1037/pha0000612. Epub 2022 Nov 10. PMID 36355684
- [Derived] Pericot-Valverde I, Heo M, Litwin AH, Niu J, Gaalema DE. Modeling the effect of stress on vaping behavior among young adults: A randomized cross-over pilot study. Drug Alcohol Depend. 2021 Aug 1;225:108798. doi: 10.1016/j.drugalcdep.2021.108798. Epub 2021 May 30. PMID 34091155